CLINICAL TRIAL: NCT04891107
Title: Feasibility and Preliminary Effects of Using a Music-based, Rhythm-modulating Wearable Sensor System in the Community in Persons With Parkinson Disease
Brief Title: Feasibility and Preliminary Effects of MR-005 in Persons With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedRhythms, Inc. (Industry)
Collaborators: Johns Hopkins University (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082000501
Record Dates: First submitted 2021-04-28; First posted 2021-05-18 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Walking Program with a Music-based, Rhythm-modulating Wearable Sensor System (Experimental)
  Interventions: Device: Walking Program with a Music-based, Rhythm-modulating Wearable Sensor System

INTERVENTIONS:
Device: Walking Program with a Music-based, Rhythm-modulating Wearable Sensor System — Participants will walk using the music-based, rhythm-modulating wearable sensor system (foot sensors, mobile device with mobile app and headphones) for thirty (30) minutes at a time, 5 times a week for 4 weeks.
  Other Names: MedRhythms MR-005 Device

SUMMARY:
The purpose of this clinical study is to evaluate the effects of music, tailored to the participant's cadence, on adherence, quality of life, gait speed, functional mobility, and walking activity in individuals with Parkinson disease when used in the home and community environment.

DETAILED DESCRIPTION:
Persons with Parkinson disease will be enrolled to determine the effects of a community walking program with a music-based device on adherence, quality of life, walking speed and walking activity. The walking program will be carried out independently by participants in their home/community environment. Noninvasive functional assessments commonly administered in clinical practice will be used to measure the variables of interest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic, typical Parkinson disease.
* Modified Hoehn and Yahr stages 1-3 per physical exam.
* Able to walk independently without physical assistance or an assistive device.

Exclusion Criteria:

* Diagnosis of atypical Parkinsonism.
* Moderately or significantly disturbing freezing episodes during daily walking.
* Cognitive impairment as determined by the Montreal Cognitive Assessment (MoCA).
* Significant hearing impairment.
* Currently participating in physical therapy.
* Cardiac problems that interfere with the ability to safely exercise.
* Orthopedic problems in the lower extremities or spine that may limit walking distance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ellis, PT, Ph.D., Principal Investigator — College of Health & Rehabilitation Sciences: Sargent College; Alex Pantelyat, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University College of Health & Rehabilitation: Sargent College, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zajac JA, Porciuncula F, Cavanaugh JT, McGregor C, Harris BA, Smayda KE, Awad LN, Pantelyat A, Ellis TD. Feasibility and Proof-of-Concept of Delivering an Autonomous Music-Based Digital Walking Intervention to Persons with Parkinson's Disease in a Naturalistic Setting. J Parkinsons Dis. 2023;13(7):1253-1265. doi: 10.3233/JPD-230169. PMID 37840504

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional participants were enrolled to account for possible attrition.
Groups:
- Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System: Will walk for 30 minutes at a time, 5 times a week, for 4 weeks using the wearable sensor system at home or in the community.
  Walking Program with a Music-based, Rhythm-modulating Wearable Sensor System: Participants will walk using the music-based, rhythm-modulating wearable sensor system (foot sensors, mobile device with mobile app and headphones) for thirty (30) minutes at a time, 5 times a week for 4 weeks.
Period: Overall Study
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Started | 26
Completed | 23
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screen failure after consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.91 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Observed Adherence (Feasibility) to Walking Program Schedule Based on Percentage of Scheduled Sessions Completed
Description: Percentage of scheduled sessions completed (5 times per week for 4 weeks)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percent of sessions completed
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 23
percent of sessions completed | 86.08696 (16.02246)

2. Primary Outcome: Safety (Feasibility) Based on the Number of Adverse Events During Training
Description: Safety as assessed by number of adverse events during training with the music-based device
Time Frame: 28 days
Measure: Number; unit: adverse events
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 23
adverse events | 0

3. Primary Outcome: Usability (Feasibility) Based on Participant Ratings on Acceptability and Usability Questionnaire.
Description: Usability as assessed by participant ratings on Acceptability and Usability Questionnaire. The Questionnaire is comprised of adapted items from the System Usability Scale, Post Study System Usability Questionnaire, Technology Assessment Model Measurement Scales, and Usefulness, Satisfaction, and Ease questionnaire as described in Ben-Zeev D, et al., 2014. Participants were asked to rate their agreement with a series of statements about the intervention (26-items) using three Likert Scale responses (disagree, neutral, or agree) for each item. The number of responses in each category of disagree, neutral, or agree were summed and averaged across the total number of participants who responded to report an overall percentage within each category of disagree, neutral, or agree on the acceptability and usability of the device. A higher overall percentage of 'agree' responses indicate a higher degree of usability as rated by participants.
Time Frame: 28 days
Measure: Number; unit: percentage of responses in a category
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 21
percentage of responses in a category
  Disagree | 21.06
  Neutral | 13.37
  Agree | 65.57

4. Primary Outcome: Change in Mobility Impact Based on the Mobility Dimension of the Parkinson's Disease Questionnaire-39 (PDQ-39) Between Baseline to Last Visit
Description: Mobility impact as assessed by Parkinson's Disease Questionnaire-39 (PDQ-39) mobility dimension (questions #1-10 from the total PDQ-39 questionnaire). Each question is scored on a 0-4 ordinal scoring system then summed to generate the sub-scale score of the mobility dimension. Lower scores represent better quality of life.
  Mobility Dimension Subscale Range: 0-100
Time Frame: 28 days
Population: Data for analysis was only obtained from 21 participants due to procedural error in instructions/administration of the test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 21
score on a scale | -1.81 (7.61)

5. Secondary Outcome: Change in Disease Severity Based on the Movement Disorders Society Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS III)
Description: Change in disease severity at baseline as compared to end of study participation (or earlier if study participant withdraws) as determined by the MDS-UPDRS III. Scores range between 0-132 with lower scores represent less disease severity.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 23
score on a scale | -3.67 (5.89)

6. Secondary Outcome: Change in Walking Endurance (m)
Description: Change in walking endurance (m) at baseline as compared to end of study participation (or earlier if study participant withdraws) as determined by the 6 Minute Walk Test (6MWT)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 23
meters | 13.83 (29.43)

7. Secondary Outcome: Change in Fast Walking Gait Speed (m/s)
Description: Change in fast walking gait speed (m/s) at baseline as compared to end of study participation (or earlier if study participant withdraws) as determined by the 10 Meter Walk Test (10MWT)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 21
meters per second | 0.001 (0.17)

8. Secondary Outcome: Overall Quality of Life Impact Based on the Total Parkinson's Disease Questionnaire -39 (PDQ-39)
Description: Overall quality of life impact at baseline as compared to end of study participation (or earlier if study participant withdraws) as assessed by Parkinson's Disease Questionnaire-39 (PDQ-39). The PDQ-39 contains 8 dimensions of function and well-being which are summed to generate the total PDQ-39 score (ranging from 0-100) where lower scores represent better quality of life.
Time Frame: 28 days
Population: Data from only 21 participants was available for analysis due to procedural error in instructions/administration of test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 21
score on a scale | -2.68 (5.14)

9. Secondary Outcome: Change in Mobility
Description: Change in mobility as measured by the Five Times Sit to Stand Test
Time Frame: 28 days
Population: Data for analysis was available for 20 participants due to due to participant inability to to perform test, therefore there was no compare functional mobility pre- and post-intervention.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 20
seconds | -1.46 (1.73)

10. Secondary Outcome: Change in Amount of Walking (Steps/Day)
Description: Change in amount (steps/day) of walking activity (proof-of-concept) at baseline as compared to during training as measured by the StepWatch Activity Monitor (SAM)
Time Frame: 8 days
Population: Data analysis available for 16 participants. Seven (7) participants had no SAM baseline data, therefore the study team could not analyze walking amount pre- and post-intervention for this measure for those participants.
Measure: Mean (Standard Deviation); unit: daily steps
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 16
daily steps | 3484 (4663)

11. Secondary Outcome: Change in Intensity (Moderate Intensity Minutes; >100 Steps/Min)
Description: Change in intensity (moderate intensity minutes; >100 steps/min) of walking activity (proof-of-concept) at baseline as compared to during training as measured by the StepWatch Activity Monitor (SAM)
Time Frame: 8 days
Population: Data analysis is available for 16 participants. Seven (7) participants did not have baseline SAM data available, therefore the study team could not analyze pre- and post-intervention changes in moderate intensity minutes for these participants.
Measure: Mean (Standard Deviation); unit: moderate intensity minutes
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
Number analyzed (Participants) | 16
moderate intensity minutes | 21.44 (23.11)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Walking Program With a Music-based, Rhythm-modulating Wearable Sensor System
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
Sample size was small and consisted of highly educated, relatively active person with mild to moderate disease severity, potentially limiting generalizability to a less active PD population with greater disease severity. The study duration of 4 weeks was relatively short and lacked a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT04891107/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT04891107/SAP_003.pdf